CLINICAL TRIAL: NCT03925753
Title: Correlation Between Autophagy-related Proteins in Peripheral Blood Mononuclear Cells and Inflammatory Markers in Hemodialysis Patients
Brief Title: Correlation Between Autophagy-related Proteins and Inflammatory Markers in Hemodialysis Patients
Status: Completed | Type: Observational
Sponsor: Tungs' Taichung Metroharbour Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 107054
Record Dates: First submitted 2019-04-22; First posted 2019-04-24 (Actual); Last update posted 2021-02-01 (Actual); Status verified 2021-01

CONDITIONS: Autophagy
Keywords: autophagy; inflammatory markers

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
One recent study demonstrated impaired autophagy in patients receiving hemodialysis (HD). To clarify whether this alteration is related to the inflammatory state in HD patients, we focused on basal autophagy in peripheral blood mononuclear cells (PBMCs) of HD patients with and without inflammation and controls. PBMCs were harvested using Ficoll density gradient centrifugation . Levels of the autophagy-associated proteins ubiquitin-binding protein p62 (p62), microtubule-associated proteins 1A/1B light chain 3A (LC3I/II) and beclin-1 in PBMCs will be detected by western blotting. Enzyme-linked immunosorbent assay kits will be used to detect the serum concentrations of interleukin (IL)-6, liposaccharide-binding protein (LBP) and tumor necrosis factor (TNF)-α.

DETAILED DESCRIPTION:
Study Design and Population

Study Design We shall enroll 30 healthy volunteers as the control group. 180 sex- and age-matched hemodialysis patients will be enrolled in this study. To be included in the study, patients have to be at least 20-years-old and on outpatient hemodialysis (HD) for at least 3 months. Patients are excluded if they had malignancy, severe liver disease (bilirubin >1.6 mg/dl), uncontrolled hypertension, severe obesity (BMI >35), currently on carbamazepine, statins or immunosuppressive agents. The medical record is thoroughly reviewed for each subject by a collaborating physician in the study. All subjects will provide written informed consent to participate and the protocol will be send to the institutional review boards of Tungs' Taichung Metroharbour Hospital

Study Parameters Predialysis blood samples are obtained on a mid-week day. Within 30 min after sampling, the remaining blood is centrifuged at 3,000 g for 10 min, immediately aliquoted and frozen at -80°C until further analysis.

Cytokine assays The following markers of inflammation and hemostasis are determined by ELISA in patients' sera: interleukin-6 (Quantikine, R&D Systems,) and plasma concentrations of CRP in a highly sensitive assay (hsCRP).

Analysis of lipids/lipoproteins Total cholesterol, highdensity lipoprotein (HDL) cholesterol, and triglyceride concentrations are determined enzymatically. Plasma glucose is measured by a glucose-oxidase method.

Measurements of Liposaccharide-binding protein (LBP) The LBP was determined from serum samples and controls using standardized enzymelinked immunosorbent assay (ELISA) methods, and serum from normal control subjects was used for interassay variation.

Isolation of PBMCs Ethylenediamine tetraacetic acid Vacutainer™ tubes are used to collect venous blood samples (10 ml) from fasting participants in the early morning. Aliquots of the supernatant are collected by centrifugation at 800 x g and 25˚C for 15 min and subsequently store at -80˚C. The remaining blood is mixed and add slowly dropwise to a centrifuge tube containing 10 ml of Ficoll separation medium. PBMCs are isolated according to manufacturer's protocol and store at -80˚C.

Western blotting PBMCs are lysed with RIPA lysis buffer and protein concentrations determined with the BCA Protein Assay kit according to the manufacturer's protocol. Subsequently, 20 μg of protein/well are separated using 12% SDS-PAGE. The proteins are subsequently transferred to nitrocellulose membranes at 300 mA for 60 min. The nitrocellulose membranes are blocked with Tris-buffered saline containing 0.1% Tween 20 (TBST) and 5% non-fat milk powder for 2 h at room temperature. The nitrocellulose membranes are incubated with primary antibodies overnight at 4˚C on a shaker set at a slow speed. The nitrocellulose membranes are washed thrice with TBST and incubated with secondary antibodies for 1 h at room temperature. After washing thrice, ECL substrate is added to the nitrocellulose membrane. The signal is detected using Image Lab™ software and band density will be quantified with imager software .

The primary antibodies against microtubule-associated proteins 1A/1B light chain 3A , ubiquitin-binding protein p62 and beclin-1 as well as GAPDH will be purchased. Peroxidase-conjugated goat anti-mouse and goat anti-rabbit secondary antibodies are used.

ELIGIBILITY:
Inclusion Criteria:

* Both sexes aged between 20-90 years.
* Received stable hemodialysis at least 3 months.
* Written informed consent.

Exclusion Criteria:

* patients with severe infections, severe heart disease and liver disease, malignancy, autoimmune disorders, severe malnutrition, or clinical conditions requiring oral nutrition supplements;
* Inability to follow protocol.
* Pregnancy or wishing/trying to get pregnant

Ages: 20 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: patients have to be at least 20-years-old and on outpatient hemodialysis (HD) for at least 3 months.
Sampling Method: Probability Sample
Enrollment: 62 (Actual)
Dates: Start 2019-03-01 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
Levels of the autophagy-associated proteins ubiquitin-binding protein p62 (p62) | 1 years
  ubiquitin-binding protein p62 (p62) in PBMCs will be detected by western blotting.
Levels of the autophagy-associated proteins microtubule-associated proteins 1A/1B light chain 3A (LC3I/II) | 1 years
  microtubule-associated proteins 1A/1B light in PBMCs will be detected by western blotting.
Levels of the autophagy-associated proteins beclin-1 | 1 years
  beclin-1 in PBMCs will be detected by western blotting.

SECONDARY OUTCOMES:
Analysis of biomarkers of Liposaccharide-binding protein (LBP) | 1 years
  The LBP was determined from serum samples and controls using standardized enzymelinked immunosorbent assay (ELISA) methods
Analysis of biomarkers of IL-6 | 1 years
  The IL-6 was determined from serum samples and controls using standardized enzymelinked immunosorbent assay (ELISA) methods was determined from serum samples and controls using standardized enzymelinked immunosorbent assay (ELISA) methods
Measurements of TNF-α | 1 years
  The TNF-α was determined from serum samples and controls using standardized enzymelinked immunosorbent assay (ELISA) methods

CONTACTS AND LOCATIONS:
Overall Officials: Paik Seong Lim, PhD, Study Chair — Tungs' Taichung Metroharbour Hospital
Locations (1):
- Tungs' Taichung MetroHarbour Hospital, Taichung, Taiwan